CLINICAL TRIAL: NCT07372898
Title: Impact of the Hospital to Home: Optimizing Preterm Infant Environment (H-HOPE) Intervention on Infants With Congenital Defects Requiring Neonatal Surgery and Their Parents.
Brief Title: Impact of Hospital to Home: Optimizing Preterm Infant Environment for Surgical Neonates and Their Parents (H-HOPE)
Acronym: H-HOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Susan Horner, PhD, Nurse Scientist, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000204
Record Dates: First submitted 2025-09-29; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Oral Feeding Outcomes; Neurodevelopment Outcome
Keywords: H-HOPE; Infant; Surgical; Congenital defect; Neonatal intensive care
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Intervention Model Description: Conceptual model: H-HOPE and Parent-Infant Outcomes Challenges faced by parents and their infants born with a congenital defect can be addressed via interventions that target early relational health. Pre-existing parental and infant biologic and social factors are known to influence the infant, parent, and parent-infant relationship. The H-HOPE intervention improves infant behavior, feeding, growth, and neurodevelopment. Mothers providing Massage+, included in the H-HOPE intervention, for their infants, report improved mental health and parenting confidence. Additionally, mothers and infants have improved neuroendocrine function, which may improve mother-infant interaction and neurodevelopment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H-HOPE (Experimental): The H-HOPE (Hospital to Home: Optimizing Preterm Infant Environment) intervention is a multisensory behavioral intervention. H-HOPE has two components: Parents+ and Massage+. Parents+: Trained study team members will provide Parents+ training using participatory guidance and experiential learning approaches. During the Parents+ sessions, parents learn infant behavioral cues, and how to read, interpret, and respond to their infant's cues during Massage+. They also learn the Massage+ intervention.
  Massage+ is a 15-minute, multisensory, behavioral intervention taught during Parents+ sessions and implemented by parents with infants in the intervention group 2x/day. It includes talking to the baby (30 seconds), massaging the baby (10 minutes; may be adapted to avoid wounds or as tolerated by baby), visual and vestibular stimuli (rocking and showing face for 5 minutes).
  Parent training will be reinforced regularly.
  Interventions: Behavioral: H-HOPE
- Control (No Intervention): Control group infants will receive ICU standard care that may include nursing care every 1-4 hours, developmental or rehabilitative therapies, parent presence, parental holding, skin-to-skin care, or other forms of infant massage. Control group parents will be offered an infant care class unrelated to the study that will include information about infant vision and hearing, sleep, and movement. Professional staff will be educated to not provide Massage+ for Control group infants. This will be reinforced with the staff and monitored daily for each patient enrolled.

INTERVENTIONS:
Behavioral: H-HOPE — The H-HOPE (Hospital to Home: Optimizing Preterm Infant Environment) intervention is a multisensory behavioral intervention. H-HOPE has two components: Parents+ and Massage+ (see Training Manual in Documents).
  Parents+: Trained study team members will provide Parents+ training using participatory guidance and experiential learning approaches. During the Parents+ sessions, parents learn infant behavioral cues, and how to read, interpret, and respond to their infant's cues during Massage+. They also learn the Massage+ intervention.
  Massage+ is a 15-minute, multisensory, behavioral intervention that will be taught to parents during Parents+ sessions and implemented by parents with infants in the experimental group. It includes talking to the baby (30 seconds), massaging the baby (10 minutes; may be adapted to avoid wounds or as tolerated by baby), visual and vestibular stimuli (rocking and showing face for 5 minutes). Trained staff may provide Massage+ when parents are not available.
  Arms: H-HOPE

SUMMARY:
Infants born with congenital defects may require major surgery in the neonatal period. These infants are at risk for neurodevelopmental impairments. Additionally, their parents are at higher risk for adverse mental health outcomes.

Early relationships are essential to healthy growth and development in all children. Relationships between parents and infants born with a congenital defect are negatively impacted by separation due to hospitalization; parental and infant stress exposures; and alterations in infant behavior and parental mental health. Benefits of H-HOPE intervention on infant neurodevelopment outcomes have been observed in healthy and at-risk term and preterm infant populations but never evaluated in infants with congenital defects. The purpose of this study is to examine impact of the Hospital to Home: Optimizing Preterm Infant Environment (H-HOPE) intervention versus standard ICU care for infants born with a congenital defect requiring neonatal surgery, and their parents. The main questions to be answered include:

1. Does H-HOPE improve pre-feeding state and behavior, oral feeding progression, and growth in infants born with a congenital defect requiring neonatal surgery?
2. Does H-HOPE neurodevelopmental outcomes in infants born with a congenital defect requiring neonatal surgery?
3. Does H-HOPE improve parental mental health outcomes among parents of infants born with a congenital defect requiring neonatal surgery?
4. Does H-HOPE improve parent-infant interactions among infants born with a congenital defect requiring neonatal surgery and their parents?
5. Does H-HOPE improve neuroendocrine function among infants born with a congenital defect requiring neonatal surgery and their parents?
6. Do parents of infants born with congenital defects requiring surgery experience participating in the H-HOPE intervention positively?

Results of this study may provide preliminary evidence supporting use of H-HOPE to positively impact short- and long-term outcomes for these infants and their parents.

DETAILED DESCRIPTION:
Primary Objectives: Primary objective of this study is to examine impact of H-HOPE intervention versus standard ICU care on early feeding, growth and neurodevelopment for infants born with a congenital defect requiring major surgery. Hypotheses include:

H1. Infants born with a congenital defect and receiving H-HOPE intervention versus standard care will have more favorable outcomes at ICU discharge and at 3-4 months including:

H1.1 Improved behavioral organization, measured by pre-feeding state and behavioral cues.

H1.2 Improved neuroendocrine function measured by salivary cortisol reactivity. H1.3 More rapid oral feeding progression and growth. H1.4 Improved neurodevelopment, measured by Test of Infant Motor Performance, Ages and Stages Questionnaire, and Parent Report of Oral Feeding at Home survey.

Secondary Objectives: Secondary objectives of study are to evaluate impact of H-HOPE intervention on parents' mental health, parents' neuroendocrine outcomes at ICU discharge, and parent-infant interactions among parents of infants born with a congenital defect requiring surgery. Secondary objectives include exploring potential relationships between parental living conditions and parent-infant outcomes related to H-HOPE. Hypotheses include:

H2. Having received H-HOPE intervention, parents of infants born with a congenital defect will have more favorable outcomes, including:

H2.1 Improved mental health, measured by perinatal depression, anxiety, and confidence in caregiving scores at ICU discharge, and perinatal PTSD at 3-4 months.

H2.2 Improved neuroendocrine function measured by salivary cortisol reactivity. H3. Having received H-HOPE intervention, parent and infant dyads will have more favorable parent-infant interactions during feeding at ICU discharge.

H 3.1 Having received H-HOPE intervention, parents will describe positive impacts of intervention on their relationship with the infant.

Background: Worldwide an estimated 6% of infants are born with a congenital defect. Congenital defects are structural anomalies that develop prenatally. These defects represent a significant cause of illness, disability, and death among children. Infants born with congenital defects, including congenital heart defects, often require specialized care in intensive care units (ICUs) and major surgery in the neonatal period. US families and the nation share the burden of costs associated with congenital defects that are estimated to be $2.6 billion per year in hospital costs alone. Throughout this application the term congenital defects refers to neonates with a birth defect requiring major surgery.

Because significant risks for neurodevelopmental impairments occur in infants with both cardiac and non-cardiac congenital defects, studies focusing on improving their neurodevelopmental outcomes are imperative. Early neurodevelopmental impairments in infants with congenital defects include difficulties with behavioral organization, oral feeding, and growth, delaying hospital progression. Significant numbers of infants with complex CHD will have neurodevelopmental impairments that frequently persist into adolescence and adulthood, including delays in cognitive, motor and language development and psychosocial issues. Cognitive, motor and language delays are observed in 23-25% of one- to three-year-old infants with non-cardiac congenital defects requiring neonatal surgery.

Parents of infants born with congenital defects experience higher risks for adverse mental health outcomes, including anxiety, depression, symptoms of trauma and post-traumatic stress disorder (PTSD). In the weeks to months following neonatal surgery to correct CHDs, 25-50% of parents report symptoms of depression and/or anxiety, 11-68% report symptoms consistent with PTSD, and 30-80% report severe psychological distress. These mental health issues may be precipitated by parental stress and grief that are triggered by the infant's diagnosis, the need for early surgery and hospitalization, and the loss of expected parenting experiences. Alterations in early parent-child relationships associated with parental mental health issues may significantly compromise parent and infant outcomes.

Frequent, repeated exposures to pain and stress impact neuroendocrine function of infants with congenital defects. Chronic activation of the hypothalamic-pituitary-adrenal axis that is associated with these cumulative exposures may alter baseline infant cortisol levels and cortisol reactivity. Stress can precipitate changes in brain structure and function that are associated with short- and long-term neurodevelopmental impairments.

Parents of infants requiring surgery to repair a congenital defect during the neonatal period experience higher levels of stress than parents of healthy infants. These may result in psychological and physiologic stress responses. Elevated cortisol in parents during the post-surgical period is associated with symptoms of post-traumatic stress at 3 months post discharge.

Quality of parent-infant interactions influences secure attachment that positively impacts later cognitive, language and social development. Parents and infants born with congenital defects are at risk for developing maladaptive interactive patterns. Parental and infant factors influence the maladaptive interaction patterns observed in this population and contribute to long term outcomes.

The Ecobiodevelopmental model explains that early experiences in a child's ecology (social and physical environment) are embedded in their biology, influencing neurodevelopment and health across the lifespan. Early relational health in the form of safe, stable, nurturing relationships are essential to healthy growth and development in all children. Unfortunately, relationships between parents and infants born with a congenital defect are negatively impacted by parental living conditions; separation due to hospitalization; parental and infant stress exposures; and alterations in infant behavior and parental mental health. There is a need for evidence-based interventions targeting early relational health in this population, and studies examining potential interventions targeting both infants and parents should be prioritized.

Parent-infant challenges faced by parents and their infants born with a congenital defect can be addressed via interventions that target early relational health. Predominantly studied with preterm infants, the H-HOPE intervention is a multisensory behavioral intervention that supports optimal infant development, parent mental health, parent-infant interactions, and stress reactivity. H-HOPE has two components: Parents+ and Massage+. Trained clinicians provide Parents+ using participatory guidance and experiential learning approaches. During the Parents+ sessions, parents learn infant behavioral cues, and how to read, interpret, and respond to their infant's cues during Massage+. They also learn the Massage+ intervention, which includes the behaviors that parents typically engage in with their infants (auditory, tactile, visual, and vestibular stimuli). After the first Parents+ session, parents begin offering Massage+ to their infants up to two times per day. While administering Massage+, parents assess their infant's behavioral cues and modify their behavior to optimize the infant's behavioral and physiologic responses. Thus, the H-HOPE intervention supports parental engagement and parent-infant interactions with hospitalized infants as parents learn about their infants' behavioral capacity. The H-HOPE intervention has not been implemented in infants born with congenital defects and their parents. This study may add to the existing knowledge related to H-HOPE.

Number of Participants: Forty total infants and one or both of their parents will be enrolled in the study. They will be randomly assigned to receive H-HOPE intervention (N=20) or standard ICU care (N=20).

Study Intervention: H-HOPE (Hospital to Home: Optimizing Preterm Infant Environment) intervention is a multisensory behavioral intervention. H-HOPE has two components: Parents+ and Massage+.

Parents+: Trained study team members will provide Parents+ training. During the Parents+ sessions, parents learn infant behavioral cues, and how to read, interpret, and respond to their infant's cues during Massage+. They also learn the Massage+ intervention.

Massage+: A 15-minute, multisensory, behavioral intervention that will be taught to parents during Parents+ sessions and implemented by parents with infants in the intervention group. It includes talking to the baby (30 seconds), massaging the baby (10 minutes; may be adapted to avoid wounds or as tolerated by baby), visual and vestibular stimuli (rocking and showing face for 5 minutes).

Parent training will be reinforced regularly. After the infant meets inclusion criteria and parents complete their Parents+ session, parents will begin offering Massage+ to their infants up to 2 times per day. While administering Massage+, parents assess their infant's behavioral cues, modifying as needed to optimize the infant's responses. Bedside nurses, child life specialists and rehabilitative therapists will be trained to provide Massage+ when a parent temporarily cannot be at the bedside (i.e., due to a sibling illness).

Control group infants will receive ICU standard care that may include nursing care every 1-4 hours, developmental or rehabilitative therapies, parent presence, parental holding, skin-to-skin care, or other forms of infant massage. Control group parents will be offered an infant care class unrelated to the study that will include information about infant sleep, and movement. Professional staff will be educated to not provide Massage+ for Control group infants. This will be reinforced with the staff and monitored daily for each patient enrolled.

Study Procedures: A randomized clinical trial will be conducted. Study procedures are outlined below. Study enrollment may occur when infant is weaning respiratory support and IV pain medications. Once enrolled, families will be randomized to intervention or control groups. Intervention group parents will not participate in Parents+ training but will be offered an infant class unrelated to study intervention.

Once enrolled infants are on respiratory support that is < a nasal cannula at 2 liters and off IV pain medications, intervention group parents will begin providing the Massage+ intervention for their infants 2 times per day, as tolerated. Parents may stop or adjust Massage+ as needed. Control group infants will receive standard ICU care, including standard parent participation activities (holding, skin-to-skin). A bedside study log will be used to document frequency of Massage+ by parents or staff, infant tolerance of Massage+ (intervention group), parent presence, and parent-infant activities for both groups. A general infant care class will also be offered to control parents.

Outcomes measures will be completed at ICU discharge and at post-ICU discharge at 3-4 months post-menstrual age.

ELIGIBILITY:
Inclusion criteria:

* Infants and one or both of their parents, born with a congenital defect and requiring major surgery during the neonatal period, including congenital heart disease.
* At the time of H-HOPE initiation, infants must be <48 weeks post-menstrual age (PMA), clinically stable (no vital sign instability during routine nursing care) on respiratory support < a nasal cannula at 2 liters per minute, and off all intravenous (IV) pain medications.

Exclusion criteria:

* Infants born at <34 weeks gestation,
* Infants born with congenital defects involving the nervous system (i.e., spina bifida, congenital hydrocephalus),
* Infants with genetic syndromes,
* Infants with a history of Extracorporeal Membrane Oxygenation,
* Infants with a history of mechanical ventilation lasting 30 or more days, or
* Infants that are wards of the state.

Ages: 1 Week to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Infant pre-feeding behavioral state | At completion of intervention period, an average of 4 weeks
  Pre-feeding state observed by trained observers in feeding video. One pre-feeding behavioral state will be assigned using the following scale 1) Quiet sleep, 2) Active sleep, 3) Drowsy, 4) Quiet alert, 5) Active alert, or 6) Crying.
Infant pre-feeding behavioral cues | At completion of intervention period, an average of 4 weeks
  Pre-feeding behavioral cues observed by trained observers in feeding video. Trained observer to record feeding readiness cues observed.
Infant oral feeding progression | Through completion of intervention period, an average of 4 weeks
  Percent of ordered feeding volume taken by mouth each day of the study
Infant growth | Through completion of intervention period, an average of 4 weeks
  Measured in grams per day of weight gain .
Infant neuroendocrine function | At completion of intervention period, an average of 4 weeks
  Infant salivary cortisol reactivity, measured immediately prior to and after receiving Massage+ with enrolled parent, or being held for 15 minutes by parent if in control group
Infant motor development | At completion of intervention period, an average of 4 weeks.
  Infant score on Test of Infant Motor Performance (TIMP). Raw scores range from 0-142, with higher scores indicative of better motor function.
Infant gross motor, fine motor, communication, problem solving, personal-social neurodevelopment | At 3-4 months infant post-menstrual age
  Infant score on Ages and Stages-3 for 3-4 month old infant; Scores range from 0-300 with higher scores indicative of better neurodevelopment
Infant feeding outcomes at home | At 3-4 month infant post-menstrual age
  Study specific survey; no numerical score but numbers of feeding problems reported will be used.

SECONDARY OUTCOMES:
Parental perinatal depression | At completion of the intervention period, an average of 4 weeks
  Perinatal depression measured using the Center for Epidemiologic Studies Depression Scale (CES-D); scores 0-60; higher score indicates more perinatal depression
Parental anxiety | At completion of intervention period, an average of 4 weeks
  Parental anxiety measured using the Child Health Worry Scale; scores 5-25; higher scale indicates more worry or anxiety about child health
Parenting confidence | At completion of intervention period, an average of 4 weeks
  Parental confidence as measured using the Karitane Parenting Confidence Scale; scores 0-45; higher scores indicate higher parental confidence.
Perinatal post-traumatic distress syndrome | At 3-4 months infant postmenstrual age.
  Score on Perinatal Post-Traumatic Stress Disorder Questionnaire-II (PPQ-II) survey; possible scores 0-13; higher score indicates increase in Perinatal PTSD
Parental salivary cortisol reactivity | At completion of intervention period, an average of 4 weeks
  Parental salivary cortisol reactivity measure before and immediately after Massage+ intervention or parent holding baby for 15 minutes (control group)
Parent-infant interactions during feeding | At completion of intervention period, an average of 4 weeks
  Measured by trained observers using the Nursing Child Assessment Satellite Training Feeding Scale; possible scores range from 0-76; increased score indicates improved interactions.
Qualitative description of H-HOPE impact on parents' relationship with their infant. | At completion of intervention period, an average of 4 weeks through 4 months infant postmenstrual age
  As measured via qualitative analysis of parent interviews with subsample of experimental group parents.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Horner, PhD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
This is a single site pilot study

REFERENCES:
- [Background] White-Traut R, Gralton K, Schmitt M, Brandon D, Kavanaugh K, Norr KF. Parents+: An Early Behavioral Intervention as a Pathway for Parent-Partnered Care. Adv Neonatal Care. 2025 Oct 1;25(5):432-440. doi: 10.1097/ANC.0000000000001288. Epub 2025 Sep 23. PMID 41020674
- [Background] White-Traut R, Brandon D, Kavanaugh K, Gralton K, Pan W, Myers ER, Andrews B, Msall M, Norr KF. Protocol for implementation of an evidence based parentally administered intervention for preterm infants. BMC Pediatr. 2021 Mar 24;21(1):142. doi: 10.1186/s12887-021-02596-1. PMID 33761902